CLINICAL TRIAL: NCT03859232
Title: Effectiveness of Cotton vs. Waterproof Cast Padding After Application of Hip Spica: A Randomized Controlled Study
Brief Title: Effectiveness of Cotton vs. Waterproof Cast Padding
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not enroll participants
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Scott Rosenfeld, Associate Professor of Orthopaedic Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-41712
Record Dates: First submitted 2018-05-30; First posted 2019-03-01 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delta Dry® Pantaloon Group (Experimental)
  Interventions: Other: Delta Dry® Waterproof Pantaloon
- Cotton Padding Group (Active Comparator)
  Interventions: Other: Cotton Padding

INTERVENTIONS:
Other: Delta Dry® Waterproof Pantaloon — Cast with newer waterproof material developed to reduce the skin complications associated with traditional cotton liners.
  Arms: Delta Dry® Pantaloon Group
Other: Cotton Padding — Cast with traditional cotton liner.
  Arms: Cotton Padding Group

SUMMARY:
This study aims to: 1) investigate the effectiveness of waterproof spica cast using Delta-Dry® Pantaloon and cast padding (BSN medical, USA) versus standard gortex pantaloon with cotton cast padding in maintaining the femur fracture and developmental dysplasia of the hip reduction after application of hip spica; 2) evaluate the overall quality ratings of both cast paddings from the perspectives of the patient and the clinicians; and 3) determine the cost difference between the both cast paddings.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients (<6 years old) diagnosed with developmental dysplasia of the hip or femur fracture who present to Texas Children's Hospital and plan to be treated with a spica cast.

Exclusion Criteria:

* Patients with thigh diameter more than 13.4 inches will be excluded because of the size limitation of the Delta-Dry Pantaloon
* Patients with femur fracture who present for treatment more than 2 weeks from the date of injury, comminuted fracture, non-displaced fracture, or with other surgical comorbidity

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2022-03-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Effectiveness as a measure of change in ratings at different time points | Baseline, 2, 6 and 12 weeks post-application
  The primary outcome (effectiveness) will be measured based on the change in ratings to the following variables/factors using a 10 point likert scale (1 being very poor and 10 being excellent):
  Comfort, Ability for the cast to dry if it became wet, Cast odor, Cast durability, Protection from skin irritation, Ease of care in the cast, Ease of Application, Padding Aesthetics, Application Time, Skin Condition, Lack of Maceration / Excoriation, Cast Odor, Padding Condition, and Ease of Removal.
  These will be collected at baseline, 2, 6 and 12 weeks post-application.

SECONDARY OUTCOMES:
Quality | Baseline, 2, 6 and 12 weeks post-application
  The secondary outcome (quality) will be measured based on rating to the following using a 10 point likert scale (1 being very poor and 10 being excellent):
  Overall Quality

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided